CLINICAL TRIAL: NCT00007956
Title: A Phase I Study Of Therapy With Mono-dgA-RFB4 In Patients With Relapsed And Refractory CD22+ B-Cell Lymphoma
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Recurrent or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068356; NCI-01-C-0021; UTSMC-99-02-07; NCT00006423 (obsolete NCT alias)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2002-02

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Biological: monoclonal antibody mono-dgA-RFB4

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have recurrent or refractory lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of monoclonal antibody mono-dgA-RFB4 in patients with recurrent or refractory B-cell lymphoma expressing CD22 antigen.
* Determine the pharmacokinetic profile of this drug in these patients.
* Correlate the pharmacokinetic parameters with the biologic effects and/or toxicity of this drug in these patients.
* Determine whether clinical responses in these patients occur at lower, equal, or higher doses than historical responses induced by a similar drug.

OUTLINE: This is a dose-escalation study. Patients are stratified according to number of circulating tumor cells in peripheral blood (more than 50/mm3 vs 50/mm3 or less).

Patients receive monoclonal antibody Mono-dgA-RFB4 IV over 4 hours on days 1, 3, and 5. Patients achieving complete, partial, or minimal remission receive additional courses of therapy every 4 weeks in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of monoclonal antibody mono-dgA-RFB4 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients achieving complete remission or stable partial remission are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or refractory B-cell lymphoma after at least 1 standard chemotherapy regimen

  * Low, intermediate, or high grade
  * CD22 antigen on at least 30% of tumor cells by flow cytometry
* No lymphoblastic lymphoma, B-cell chronic lymphocytic leukemia, B-cell or pre-B-cell acute lymphocytic leukemia, or hairy cell leukemia
* Measurable disease

  * Positive bone marrow not considered measurable
  * Circulating tumor cells in peripheral blood considered measurable
* No CNS disease (leptomeningeal or parenchymal)
* No lymphomatous or infectious pulmonary parenchymal disease
* No baseline/pleural effusion
* Ineligible for or refused autologous or allogeneic bone marrow transplantation NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count greater than 50,000/mm^3
* Absolute granulocyte count greater than 750/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGPT less than 2 times upper limit of normal
* Albumin greater than 75% lower limit of normal

Renal:

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* Ejection fraction greater than 40% by MUGA or echocardiogram

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No human anti-mouse antibody (HAMA) levels greater than 1 microgram/mL
* No condition that may require stenting of ureters, stabilization of impending pathological fractures, or relief of airway, bowel, or biliary tract obstruction
* No other concurrent illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy and recovered
* No concurrent chemotherapy

Endocrine therapy:

* No concurrent corticosteroids unless receiving stable maintenance dose prior to therapy

Radiotherapy:

* No prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: Edward A. Sausville, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Center for Cancer Research, Bethesda, Maryland